CLINICAL TRIAL: NCT04364477
Title: The Effect Of The Transversus Abdominis Plane Block On Postoperative Analgesia and Patient Comfort In Patients Having Abdominal Surgery With General Anesthesia
Brief Title: TAP Block On Abdominal Surgery Patients With General Anesthesia
Acronym: TAPBLOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Cemil Isbir, Assoc. Prof., Cumhuriyet University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Other Identifier-2018
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Post-Op Complication; Pain, Postoperative
Keywords: TAP block; postoperative pain; Bupivacaine; ultra sound guided regional anesthesia
MeSH Terms: conditions — Postoperative Complications; Pain, Postoperative | interventions — Dental Occlusion; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tap block Group (Active Comparator): Tap Block group :(Group 1) After General anestehesia At the end of the operation, TAP blocks were placed to the 1st group patients.
  Interventions: Procedure: transversus abdominis plane (TAP) block
- Control Group (Placebo Comparator): No block applied. only General anesthesia was applied.
  Interventions: Procedure: transversus abdominis plane (TAP) block

INTERVENTIONS:
Procedure: transversus abdominis plane (TAP) block — The transversus abdominis plane (TAP) block is a regional anesthesia technique described in recent years that provides analgesia for the anterior portion of the abdominal wall after abdominal surgery.
  Other Names: General Anesthesia

SUMMARY:
INTRODUCTION: The aim of this study was to investigate the effects of tranversus abdominis plane (TAP) block placed postoperatively using ultrasound guidance for patients with caesarean section, myomectomy and hysterectomy under general anesthesia by eliminating additional pain caused by surgical incision.

MATERIALS AND METHODS: The study has been planned to investigate the postoperative analgesia of 50 patients with TAP blocks applied and non-applied between the ages of 18-65, who will pass abdominal surgery. Study has been conducted in a prospective, randomized and controlled manner. Patients have been classified as those who have undergone TAP block (group: I) and those without block (group: II).

DETAILED DESCRIPTION:
The study was conducted in accordance with the Helsinki Declaration Principles (rev.2013) and with the approval of the local ethical board. After the written and signed approval of the patients, it has been planned to investigate the postoperative analgesia and comfort of a total of 50 patients The study examined the postoperative pain levels after abdominal surgery with and without TAP block. Subjects were between the ages of 18-65 who will have abdominal surgery with transverse incision (cesarean section, hysterectomy (benign), myomectomy) and American Society of Anesthesiologists Physical Status Classification System (ASA) I-II. Our study is planned to be prospective, randomized and controlled. The individuals to be engaged were divided into two groups in a randomized form. Randomization was based on a computer-generated code. In the first group, a total of 25 patients were admitted with 16 cesareans, 6 myomectomies and 3 hysterectomies applied to the TAP block. In the second group, a total of 25 patients who did not undergo TAP block, no needle intervention, 18 cesareans, 5 myomectomies and 2 hysterectomies were included as the control group. Those with skin infections, patients with organomegaly (hepatomegaly and splenomegaly), people who did not give consent to the method, and individuals with allergies to drugs to be used in the intervention area where Transversus abdominis plane is to be conducted were not included in the study.

Isolyte® balanced electrolyte solution at a rate of 2 ml/kg/hour was administered to the individuals whose oral intake was discontinued 8 hours before the surgery. The individuals to be included in the study were not given any sedative agent on the morning of their surgery. 10 cm visual analog scale (VAS) was explained in detail to all patients before the procedure. All individuals to be included in the study were followed up with anesthesia monitor (Drager Infinity Vista XL®), heart rate (CAH), electrocardiography (ECG) (lead II), systolic blood pressure (SKB) and diastolic blood pressure (DBP) in the preoperative and preoperative period. After induction of anesthesia with 1 µg/kg fentanyl (Fentanyl, Janssen-Cilag), 0.5 mg/kg rocuronium bromide (Esmeron® vial, Schering-Plough) and 5 mg/kg thiopental sodium (Pental Sodium®, I.E Ulagay), 4-6% Desflurane (Suprane® Volatile Solution, Pharmacist-Head - Baxter) and 50% N2O in Oxygen were used to maintain anesthesia following endotracheal intubation. Differently in general anesthesia management at cesarean operations, 5 mg/kg thiopental sodium (Pental Sodium®, I.E Ulagay) and 0.5 mg/kg rocuronium bromide (Esmeron® vial, Schering-Plough) were administered in induction and 4-6% Desflurane (Suprane® Volatile Solution, Pharmaceutical-headed-Baxter), (50% N2O+50% Oxygen) and 1 µg/kg fentanyl (Fentanyl, Janssen-Cilag) are added as inhalation anesthesia after umbilical cord clamping in maintenance. The maintenance dose of rocuronium bromide was 0.15 mg/kg for all cases. Necessary fluid replacement was performed during the operation. At the end of the operation, TAP blocks were placed to the 1st group patients.

After the necessary sterilization conditions were established, the linear ultrasound probe was sterilely coated and placed in the middle of the iliac crest with the end limit of the ribs. Starting with skin, the layers in descending order, subcutaneous adipose tissue, external oblique muscle, internal oblique muscle, transversus abdominis muscle and peritoneum were identified. As the tip of the 21Gx100 mm needle (Pajunk®-Uniplex Nanoline cannula with facet tip) passed through the muscular layers and fascia, a fascial click was felt and the needle was advanced with ultrasound in a controlled manner. After receiving the second click sensation (passage of the fascia of the internal oblique muscle), after a 0.5-1 ml test dose, the location of the needle was fixed and frequently aspirated and applied to the bilateral neurophysical plan so that 20 ml of 0.25% bupivacaine (Marcaine® 0.5%, Astra Zeneca) was applied to one side.

The first group of patients were awakened after TAP block treatment and reversal of muscle relaxant with atropine sulphate and neostigmine; the control group was awakened after reversal of muscle relaxant with atropine sulphate and neostigmine at the end of the operation. When VAS>3 in the postoperative period, 1g of paracetamol was administered as an intravenous infusion over 10 minutes in terms of the first analgesic requirement.

Systolic and diastolic arterial pressures, heart rate of all patients were monitored immediately before and postoperatively at 30th minute and 1st, 2nd, 4th, 6th, 12th and 24th hours after block administration. The pain levels of the patients were measured at the 30th minute, 1st, 2nd, 4th, 6th, 12th and 24th postoperative VAS values. The need for nausea, vomiting, and initial analgesia was recorded. In this study, none of the patients underwent any invasive procedures other than routine procedures.

When parametric test counts were fulfilled (Kolmogorov-Simirnov) by uploading the data obtained from our study to SPSS (ver:22.0) program, significance test of the difference between the two averages, variance analysis in repeated measurements, Bonferroni test, Mann Whitney U test, Wilcoxon test, Freidman test and Chi-square test were used when parametric test assumptions were not fulfilled. When α is taken as 0.05, β: 0.10, 1-β: 0.90, 25 individuals were included in each group and the strength of the test was p= 0.90388.

Our data were reported as arithmetic mean, standard deviation, number of individuals and the level of error was taken as 0.05.

ELIGIBILITY:
Inclusion Criteria: 1) ASA I and II patients. 2) Healthy people.

Exclusion Criteria: 1)Those with skin infections, 2) Patients with organomegaly (hepatomegaly and splenomegaly), 3) People who did not give consent to the method. 4) Individuals with allergies to drugs to be used in the intervention area where Transversus abdominis plane is to be conducted were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-04 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale of patients | 0-30 minutes
  Pain scale
Sistolic Blood Pressure of patients | 0-30 minutes
  Sistolic Blood Pressure
Need For Analgesic drugs for post-op patients | 0-60 minutes
  Analgesic need
patients with nausea | 0-60 minutes
  post op nausea

IPD SHARING:
Plan to Share IPD: No